CLINICAL TRIAL: NCT01879787
Title: Impact of Transcranial Direct Current Stimulation (tDCS)on the Effects of Mental Practice and Modified Constraint-induced Movement Therapy (mCIMT)in the Rehabilitation of Chronic Stroke Patients
Brief Title: Effects of tDCS Combined With mCIMT or Mental Practice in Poststroke Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, PhD in Neuroscience, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS_mCIMT_MP_Stroke
Record Dates: First submitted 2013-05-10; First posted 2013-06-18 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2014-05

CONDITIONS: Stroke
Keywords: Stroke; transcranial direct current stimulation; constraint-induced movement therapy; mental practice
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- physiotherapy + anodal tDCS + mCIMT (Experimental): Before a anodal tDCS with duration of 13 minutes and intensity of 1mA applied at the injured motor cortex, the patient will be submitted to a 30 minutes physiotherapy protocol. Lastly the individual will realized a 45 minutes mCIMT protocol. The experimental sessions will be repeated three times per week, will be realized 10 sessions. At home the patient will spend 6 hours per day with the restraint for the paretic upper limb.
  Interventions: Other: tDCS
- Physiotherapy + cathodal tDCS + mCIMT (Experimental): Before a cathodal tDCS with duration of 9 minutes and intensity of 1mA applied at the healthy motor cortex, the patient will be submitted to a 30 minutes physiotherapy protocol. Lastly the individual will realized a 45 minutes mCIMT protocol. The experimental sessions will be repeated three times per week, will be realized 10 sessions. At home the patient will spend 6 hours per day with the restraint for the paretic upper limb.
  Interventions: Other: tDCS
- Physiotherapy+bi-hemispheric tDCS+mCIMT (Experimental): Before a bi-hemispheric tDCS with duration of 13 minutes and intensity of 1mA applied at the healthy (cathode) and injured (anode) motor cortex, the patient will be submitted to a 30 minutes physiotherapy protocol. Lastly the individual will realized a 45 minutes mCIMT protocol. The experimental sessions will be repeated three times per week, will be realized 10 sessions. At home the patient will spend 6 hours per day with the restraint for the paretic upper limb.
  Interventions: Other: tDCS
- Physiotherapy+sham tDCS+mCIMT (Sham Comparator): Before a sham tDCS with duration of 30 seconds and intensity of 1mA applied at the injured motor cortex, the patient will be submitted to a 30 minutes physiotherapy protocol. Lastly the individual will realized a 45 minutes mCIMT protocol. The experimental sessions will be repeated three times per week, will be realized 10 sessions. At home the patient will spend 6 hours per day with the restraint for the paretic upper limb.
  Interventions: Other: tDCS
- Physiotherapy+tDCS+mental practice (Experimental): Before a tDCS protocol applied during de mental practice training , the patient will be submitted to a 30 minutes physiotherapy protocol. The experimental sessions will be repeated three times per week, will be realized 10 sessions.
  Interventions: Other: tDCS
- Physiotherapy+sham tDCS+mental practice (Sham Comparator): Before a sham tDCS protocol applied during the mental practice training, the patient will be submitted to a 30 minutes physiotherapy protocol. The experimental sessions will be repeated three times per week, will be realized 10 sessions.
  Interventions: Other: tDCS
- Physiotherapy (No Intervention): The patient will be submitted to a 30 minutes physiotherapy protocol. The experimental sessions will be repeated three times per week, will be realized 10 sessions.

INTERVENTIONS:
Other: tDCS — tDCS involves application of very low-amplitude direct currents(2 mA or less) via surface scalp electrodes.This produces a sub-sensory level of electrical stimulation which remains imperceptible by most people during its application. In a small percentage of patients it may cause minimal discomfort with a mild tingling sensation, which usually disappears after a few seconds. The applied current modifies the transmembrane neuronal potential and thus influences the level of excitability. Depending on the polarity of active electrodes tDCS can increase or decrease corticomotor excitability. Cathodal tDCS decrease and anodal tDCS increase the motor cortex excitability.
  Other Names: non invasive brain stimulation
  Arms: Physiotherapy + cathodal tDCS + mCIMT; Physiotherapy+bi-hemispheric tDCS+mCIMT; Physiotherapy+sham tDCS+mCIMT; Physiotherapy+sham tDCS+mental practice; Physiotherapy+tDCS+mental practice; physiotherapy + anodal tDCS + mCIMT

SUMMARY:
This study aims to evaluate systematically and controlled the effectiveness of mental practice techniques and modified constraint- induced movement therapy (mCIMT)in the treatment of post-stroke patients with motor deficit in the upper limb. As well as finding a protocol of transcranial direct current stimulation(tDCS)that will maximize the effects of the practice of mental image and mCIMT. To this end, the subjects included will be submitted to 12 therapy sessions with active or sham tDCS combined with at least one of the following techniques: conventional physiotherapy, mental practice technique or mCIMT

DETAILED DESCRIPTION:
Eighty-four patients chronic post-stroke will be recruited to participate in the study. After screening to check the eligibility criteria and giving informed consent, the patients will be randomized into seven distinct groups (12 per group). All the patients will be submitted to 12 therapeutic sessions that will occur with a frequency of three times a week.

Before, immediately after and 1 month after the beginning of the experimental sessions patients will be submitted to an evaluation at each moment will be applied: (i) Fugl- Meyer Scale, (ii) Motor Activity Log Scale, (iii ) Jebsen-Taylor hand functional test, (iv) Independence Functional Measure (v) Box-Block Test, (vi) Dynamometry and (vii) Berg Balance Scale.

In experimental sessions, the subjects always receive physiotherapy treatment with conventional techniques, the protocol will follow the guidelines outlined in Clinical Practice Guideline for physical therapy in stroke patients with the Royal Dutch Society for Physical Therapy (2004). Besides physical therapy, the patient may be subjected to transcranial direct current stimulation (tDCS) associated with the techniques of modified constraint-induced movement therapy (mCIMT) or mental practice (MP).

tDCS protocol During tDCS sessions, the patients will be seated in a comfortable chair with head and arm rests. Continuous direct current will be applied by clinical microcurrent stimulator (Soterix, USA) using a pair of saline-soaked surface sponge electrodes (surface 35 cm2). For anodal and sham stimulation (the polarity refers always to the motor cortical electrode), the anode electrode will be placed over primary motor cortex (M1; EEG 10/20 system) of the affected hemisphere and cathode above contralateral orbit. For cathodal tDCS, the cathode will be positioned over M1 of the non-affected hemisphere and the anode was placed above the contralateral orbit. For bi-hemispheric tDCS the anode electrode will be placed over M1 of the affected hemisphere and the cathode over the M1 of the healthy hemisphere. Transcranial direct current stimulation will be administered with a current strength of 1 mA for 13 (anodal/bi-hemispheric tDCS) or 9 min (cathodal tDCS). Sham tDCS will be performed by current flow for 30 s, a method shown to achieve a good level of blinding mCIMT protocol The modified CIMT consisted of (i) complete immobilization of the non-paretic upper limb and (ii) intensive training the paretic upper limb and will be administered by a trained therapist, who was not involved in the pre-post evaluations.

Continuously for six hours daily over a period of four weeks, including weekend, all patients will be remained with complete immobilization of the non paretic upper limb. For this, an arm sling with the shoulder in adduction and internal rotation, elbow flexed at 90º, wrist and fingers in neutral position, made specifically for each patient will be used. They will be advised to use the restriction during their daily activities and instructed to remove it every hour for 10 minutes to perform stretching, which has been previously taught by the researchers to avoid functional deterioration caused by disuse. All muscle groups of the upper extremity will be stretched. A guide with instructions of the stretching will be distributed to patients. The patients will be instructed to take the immobilization on every day at same hour the tDCS sessions. In addition, the patients will be allowed to take the arm sling off during activities in which safety would be compromised, such as toileting, dressing, and bathing.

For intensive training the paretic upper limb, the patients will attend a gross motor and fine motor activities program performed for 1 hour per day, three times per week. Each task was performed for 2-3 minutes and the rest interval between tasks will be determined for each subject in order to avoid fatigue and excessive tiredness. The tasks will be progressively adapted by increasing speed or accuracy to allow improvement of patient performance. All tasks will be done with subjects sitting on a chair with standard dimensions and performed on support table. During training sessions, the patients will remain with the non-paretic arm immobilized.

Mental practice protocol Prior to experimental sessions, the mental capacity of subjects to learn the imagery techniques will be tested by the Kinesthetic and Visual Imagery Questionnaire and a chronometric test. The Kinesthetic and Visual Imagery Questionnaire is an imagery assessment tool comprised of 10 items, each scored on a five-point ordinal scale, including the image clarity (visual dimension) and the sensations intensity (kinesthetic dimension) of body movements. Each item describes an action: (i) neck flexion/extension, (ii) shoulder shrugging, (iii) forward trunk flexion, (iv) forward shoulder flexion, (v) elbow flexion, (vi) thumb to finger tips, (vii) knee extension, (viii) hip abduction, (ix) foot external rotation, and (x) foot tapping. Subjects physically execute each movement and immediately afterwards imagine performing the same movement. A score of 5 corresponds to the highest clarity/intensity, and a score of 1 corresponds to the lowest clarity/ intensity (for a review, see Malouin et al., 2007). The Kinesthetic and Visual Imagery Questionnaire scores allowed the researcher to assess each participant's abilities and decide whether the subject was a suitable candidate for MP. Comparing actual and imagined movement times, the chronometric test determined the motor imagery ability of participants.

The mental practice will consist of motor imagination of tasks. These tasks will consist of action for the patient to imagine themselves, with the greatest wealth of detail possible, performing motor activities with the hemiparetic upper limb, such as the movement of the touching thumb on each other's toes hand, or even the movement of bringing a cup towards his mouth. The technique of mental practice will be applied at the same time of the tDCS.

ELIGIBILITY:
Inclusion Criteria:

* chronic stroke (> 6 months)
* score ≥ 20 at the Folstein Mini Mental State Examination
* score ≤ 3 at the Ashworth Scale
* score ≤ 4 at the Visual Analog Pain Scale

Exclusion Criteria:

* multiple brain lesions
* medication for treatment of spasticity
* attention deficit
* deficit in perceptual ability and motivation to follow the instructions for the mental training
* pregnant
* pacemaker
* metal implant in the region of the skull and face
* history of convulsion
* epilepsy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Fugl-Meyer Assessment of Upper Extremity Motor Function | At baseline, 1 month and 2 month
  The Fugl-Meyer assessment was used to measure recovery of motor control. It is a 226-point scoring system that includes range of motion, pain, sensation, motor function of the upper and lower extremities, and balance.This instrument provides a reliable and valid measure of specific motor function that is also sensitive to change.

SECONDARY OUTCOMES:
Change from Motor Activity Log | At baseline, 1 month and 2 month
  The MAL is a scripted, structured interview to measure real-world upper extremity function. It was developed to measure the effects of therapy on the more impaired arm following stroke. The original MAL consists of 14 activities of daily living (ADLs) such as using a towel, brushing teeth, and picking up a glass. For a specified time period post-stroke, the individual is asked about the extent of the activity performed and how well it was performed by the more impaired arm. The response scale ranges from 0 (never used) to 5 (same as pre-stroke). The mean of the scores for frequency of the activity comprises the Amount of Use (AOU) scale; the mean of the scores for how well the activity was performed comprises the Quality of Movement (QOM) scale. Ideally, ratings are obtained from the individual with a stroke as well as a knowledgeable informant (caregiver).

OTHER OUTCOMES:
Change from Jebsen-Taylor Hand Function Test | At baseline, 1 month and 2 months
  The Jebsen-Taylor function test was designed to provide a short, objective test of hand functions commonly used in activities of daily living (ADLs). The target patient population includes adults with neurological or musculoskeletal conditions involving hand disabilities, although there may be other patient populations with other hand dysfunctions which may be appropriate. The test was developed to be used by health professionals working in restoration of hand function. It consists of seven items that include a range of fine motor, weighted and non-weighted hand function activities

CONTACTS AND LOCATIONS:
Overall Officials: Kátia K Monte Silva, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil